CLINICAL TRIAL: NCT04155424
Title: A Phase 2/3 Open-Label, Single-Arm Trial to Evaluate the Safety and Activity of Eculizumab in Pediatric Patients With Relapsing Neuromyelitis Optica Spectrum Disorder
Brief Title: A Study of the Safety and Activity of Eculizumab in Pediatric Participants With Relapsing Neuromyelitis Optica Spectrum Disorder
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Pediatric clinical study is not feasible.
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECU-NMO-303; 2019-001829-26 (EudraCT Number)
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Results first posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Neuromyelitis Optica; Neuromyelitis Optica Spectrum Disorder
Keywords: Neuromyelitis Optica; Neuromyelitis Optica Spectrum Disorder; Devic's Disease; Transverse Myelitis; Optic Neuritis; Relapse; Eculizumab; Soliris; CNS Autoimmune Disorders; Demyelinating Disorders; NMO; NMOSD
MeSH Terms: conditions — Neuromyelitis Optica; Myelitis, Transverse; Optic Neuritis; Recurrence; Demyelinating Diseases | interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Eculizumab (Experimental): All participants will receive open-label eculizumab by intravenous infusion during the Primary Treatment Period, starting on Day 1 and for a total of 52/53 weeks. The dosing regimen will be based on the participant's body weight. As body weight changes during the study, the participant's weight cohort and dose may change accordingly.
  After completing the 52/53-week Primary Treatment Period, participants may continue receiving eculizumab in the Extension Treatment Period for 104 weeks.
  Interventions: Drug: Eculizumab

INTERVENTIONS:
Drug: Eculizumab — Following a weight-based weekly dose of eculizumab during an induction phase, participants will receive weight-based doses of eculizumab every 2 weeks during the Primary Treatment Period and Extension Treatment Period.
  Other Names: Soliris

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of eculizumab in pediatric participants (aged 2 to < 18 years) with relapsing neuromyelitis optica spectrum disorder (NMOSD).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged 2 years to < 18 years with body weight ≥ 10 kilograms (kg).
2. Vaccinated against Neisseria meningitidis within 3 years prior to, or at the time of initiating eculizumab. Participants who initiate study drug treatment less than 2 weeks after receiving a meningococcal vaccine must receive appropriate prophylactic antibiotics until 2 weeks after the vaccination.
3. Documented vaccination against haemophilus influenzae type b and streptococcus pneumoniae infections at least 2 weeks prior to dosing as per local and country-specific immunization guidelines for the appropriate age group.
4. Anti-aquaporin-4 antibody-positive and diagnosis of NMOSD as defined by the 2015 International Panel for Neuromyelitis Optica Diagnosis criteria.
5. Historical Relapse Rate of at least 2 relapses in the last 2 years, and with at least 1 relapse in the year prior to Screening.
6. EDSS score ≤ 7.
7. Participants who enter the study receiving supportive immunosuppressive therapies (ISTs) for the prevention of relapse, either in combination or monotherapy, must be on a stable dosing regimen of adequate duration.
8. Female participants of childbearing potential must have a negative pregnancy test (serum human chorionic gonadotropin) at Screening and follow protocol-specified contraception guidance for avoiding pregnancy while on treatment and for 5 months after the last dose of eculizumab.
9. Male participants with a female spouse/partner of childbearing potential or a pregnant or breastfeeding spouse or partner must agree to use double barrier contraception (male condom plus appropriate barrier method for the female partner) while on treatment and for at least 5 months after the last dose of eculizumab.

Exclusion Criteria:

1. Parent or legal guardian is an Alexion employee.
2. Pregnant, breastfeeding, or intending to conceive during the course of the study.
3. Participants known to be human immunodeficiency virus positive or with congenital immunodeficiency.
4. Unresolved meningococcal or other serious infection.
5. Any unresolved acute or chronic systemic bacterial or other infection that is clinically significant in the opinion of the Investigator and has not been treated with appropriate antibiotics.
6. Use of rituximab or other biologicals such as tocilizumab within 6 months prior to Screening.
7. Use of mitoxantrone within 3 months prior to Screening.
8. Use of intravenous immunoglobulin or plasma exchange within 3 weeks prior to Screening.
9. Use of immunomodulatory therapies for multiple sclerosis within 3 months prior to Screening.
10. Has previously received treatment with eculizumab or other complement inhibitors.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (35):
- United States (15):
  - Clinical Trial Site, San Francisco, California
  - Clinical Trial Site, Washington D.C., District of Columbia
  - Clinical Trial Site, Miami, Florida
  - Clinical Trial Site, Atlanta, Georgia
  - Research Site, Baltimore, Maryland
  - Clinical Trial Site, Rockville, Maryland
  - Clinical Trial Site, Boston, Massachusetts
  - Research Site, Boston, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Hackensack, New Jersey
  - Research Site, New Brunswick, New Jersey
  - Research Site, New York, New York
  - Clinical Trial Site, Chapel Hill, North Carolina
  - Clinical Trial Site, Philadelphia, Pennsylvania
  - Research Site, Dallas, Texas
- Canada (5):
  - Research Site, Calgary, Alberta
  - Clinical Trial Site, Edmonton, Alberta
  - Research Site, Toronto, Ontario
  - Clinical Trial Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- Germany (3):
  - Clinical Trial Site, Regensburger Straße, Goettingen
  - Research Site, Datteln
  - Research Site, Münster
- Italy (6):
  - Research Site, Catania
  - Research Site, Gallarate
  - Clinical Trial Site, Genoa
  - Research Site, Genova
  - Research Site, Rome
  - Clinical Trial Site, Rome
- Japan (2):
  - Research Site, Yokohama
  - Clinical Trial Site, Yokohama
- Clinical Trial Site, Seoul, South Korea
- Spain (3):
  - Clinical Trial Site, Barcelona
  - Research Site, Esplugues de Llobregat
  - Clinical Trial Site, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ECU-NMO-303&attachmentIdentifier=4f09d77b-c7f0-437d-8901-b158798b7a5c&fileName=ecu-nmo-303_CSR_Synopsis_Redcted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All 5 participants were in the >=40 kilograms (kg) weight cohort at enrollment. Therefore, all 5 participants received the same dose of study drug for the Induction Period and the Maintenance Period as described in the study arm.
Groups:
- Eculizumab: Induction Period: Participants received eculizumab (900 milligrams [mg]) via intravenous (IV) infusion once a week for 4 weeks. Maintenance Period: Participants received eculizumab (1200 mg) via IV infusion every 2 weeks from fifth dose (Week 4) onwards and then every 2 weeks.
Period: Overall Study
Arm/Group | Eculizumab
Started | 5
Received at Least 1 Dose of Study Drug | 5
Number of Participants Who Received Study Drug During the Induction Period | 5
Number of Participants Who Received Study Drug During the Maintenance Period | 5
Completed | 0
Not Completed | 5
Not completed — Other than specified | 3
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Safety Set included all participants who received at least 1 dose of eculizumab.
Groups:
- Eculizumab: Induction Period: Participants received eculizumab (900 mg) via IV infusion once a week for 4 weeks. Maintenance Period: Participants received eculizumab (1200 mg) via IV infusion every 2 weeks from fifth dose (Week 4) onwards and then every 2 weeks.
Arm/Group | Eculizumab
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.0 (4.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Change Between the Baseline Annualized Relapse Rate (ARR) and the On-Trial ARR at Week 52/53
Description: ARR was calculated as the number of relapses for each participant divided by the number of years of treatment for that participant. Baseline ARR was based on 24 months prior to screening.
Time Frame: Baseline, Week 52/53
Population: Full Analysis Set included all participants who received at least 1 dose of eculizumab. Here, overall number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: relapses per participant per year
Arm/Group | Eculizumab
Number analyzed (Participants) | 5
relapses per participant per year | -3.01 (2.504)

2. Primary Outcome: Time to First On-trial Relapse
Description: Time to First Relapse was defined as beginning at the time the participant's first dose of eculizumab was administered until the participant's first on-trial relapse was reported by the Investigator. Participants who did not experience an on-trial relapse were censored at the end of the study period.
Time Frame: Baseline up to Week 52/53
Population: Full Analysis Set included all participants who received at least 1 dose of eculizumab. Note that since no participants experienced a On-trial Relapse, data was not collected for this Outcome Measure.
Arm/Group | Eculizumab
Number analyzed (Participants) | 0

3. Secondary Outcome: Change From Baseline in Expanded Disability Status Scale (EDSS) Score at Week 52/53
Description: Disease-related disability was measured by the EDSS. The EDSS is an ordinal clinical rating scale that ranges from 0 (normal neurologic examination) to 10 (death) in half-point increments. A decrease in score indicates improvement.
Time Frame: Baseline, Week 52/53
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Eculizumab
Number analyzed (Participants) | 4
score on a scale | -0.75 (1.708)

4. Secondary Outcome: Change From Baseline in the Hauser Ambulation Index (HAI) Score at Week 52/53
Description: The HAI evaluates gait and was used to assess the time and effort used by the participant to walk 25 feet (8 meters). The scale ranged from 0 to 9, with 0 being the best score (asymptomatic; fully ambulatory with no assistance) and 9 being the worst (restricted to wheel chair; unable to transfer self independently). A decrease in score indicates improvement.
Time Frame: Baseline, Weeks 52/53
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Eculizumab
Number analyzed (Participants) | 4
score on a scale | 0.0 (0.00)

5. Secondary Outcome: Change From Baseline in Pediatric Quality of Life Inventory (PedsQL) Score at Week 52/53
Description: PedsQL included a child self-report for participants 5 to 18 years with a 23-item PedsQL Generic Core Scales report. The PedsQL Generic Core Scales report included 4 scales, physical functioning, emotional functioning, social functioning, and school functioning. Each item used a 5-point rating scale (from 0=never to 4=almost always). Items are reverse scored and linearly transformed to a 0 (almost always) -100 (never) scale. All summary/total scores were mean of specific items where higher score indicated better HRQoL.
Time Frame: Baseline, Weeks 52/53
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Eculizumab
Number analyzed (Participants) | 4
score on a scale | -5.01 (10.401)

6. Secondary Outcome: Number of Participants With Shift From Baseline in Visual Acuity (VA)
Description: The Snellen chart was used to assess VA. The Snellen chart quantifies ability to read letters of varying sizes at a fixed distance in relation to the distance at which a participant with normal vision could read the same letters. The test was performed at a standard distance, typically 6 meters or 20 feet. The Snellen chart is typically recorded as acuity ratio distance (6 meters or 20 feet), so for normal VA it would be recorded as 20/20 or 6/6. Visual acuity was summarized according to the eye with greater worsening at the end of primary treatment period (Week 52/53). Data are presented for number of participants with a shift from baseline in VA presented per the different levels of acuity ratio distance. Baseline was defined as the last available assessment prior to the first IP study drug infusion for all participants regardless of treatment group. Visual Acuity data are only reported for the categories with available data at Baseline and Week 52/53.
Time Frame: Baseline, Week 52/53
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 4
Participants
  Shift from VA 20/20-20/29 to VA 20/20-20/29 | 3
  Shift from VA 20/30-20/59 to VA 20/20-20/29 | 1

7. Secondary Outcome: Number of Participants With Shift From Baseline in Confrontational Visual Fields (VF)
Description: Confrontational visual fields were summarized according to the number of quadrants with deficits across both eyes. Baseline was defined as the last available assessment prior to the first IP study drug infusion for all participants regardless of treatment group.
Time Frame: Baseline, Weeks 52/53
Population: Full Analysis Set included all participants who received at least 1 dose of eculizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 3
Participants
  0 to 0 | 2
  2 to 0 | 1

8. Secondary Outcome: Number of Participants With Shift From Baseline in Color Vision
Description: Color vision was evaluated as the shift from baseline and described for participants with normal color vision at baseline in at least one eye. Participants with 13 or less correctly identified Ishihara plates were considered as having abnormal color vision, participants with 14 or more correctly identified plates were considered as having normal color vision. Baseline was defined as the last available assessment prior to the first IP study drug infusion for all participants regardless of treatment group.
Time Frame: Baseline, Weeks 52/53
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 4
Participants
  No Change from Normal | 4
  Worsened from Baseline | 0

9. Secondary Outcome: Serum Eculizumab Concentration at Week 52
Time Frame: Week 52
Population: Pharmacokinetic/Pharmacodynamic (PK/PD) analysis set included participants who received at least 1 dose of eculizumab and who had evaluable PK/PD data for the endpoint.
Measure: Mean (Standard Deviation); unit: micrograms/milliliters
Arm/Group | Eculizumab
Number analyzed (Participants) | 3
micrograms/milliliters
  Pre-dose: 5-90 Minutes | 460.7 (65.04)
  Post-dose: 60 minutes | 971.3 (198.04)

10. Secondary Outcome: Change From Baseline in Serum Free Complement Protein 5 (C5) Concentrations at Week 52
Time Frame: Baseline, Week 52
Population: PK/PD analysis set included participants who received at least 1 dose of eculizumab and who had evaluable PK/PD data. for the endpoint. Here, overall number of participants analyzed signifies those participants who were evaluable for this outcome measure .
Measure: Mean (Standard Deviation); unit: micrograms/milliliters
Arm/Group | Eculizumab
Number analyzed (Participants) | 3
micrograms/milliliters
  Baseline | 166.67 (50.203)
  Change from Baseline at Week 52 | -166.64 (50.194)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 53
Description: Treatment emergent adverse events (TEAEs) are AEs with a start date on or after the date of the first dose of study intervention. TEAEs were analyzed for Safety Set which included all participants who received at least 1 dose of eculizumab.
Arm/Group | Eculizumab
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eculizumab (N=5)
Liver function test increased (Investigations) | 1
Encephalitis meningococcal (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Eculizumab (N=5)
Abdominal pain lower (Gastrointestinal disorders) | 1
Bowel movement irregularity (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Feeling abnormal (General disorders) | 1
Pyrexia (General disorders) | 1
Vaccination site erythema (General disorders) | 1
Vaccination site pain (General disorders) | 1
COVID-19 (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Vulvovaginal candidiasis (Infections and infestations) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Growing pains (Musculoskeletal and connective tissue disorders) | 1
Kyphosis (Musculoskeletal and connective tissue disorders) | 1
Weight increased (Investigations) | 1
Headache (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Chalazion (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Hepatic steatosis (Hepatobiliary disorders) | 1
Post vaccination fever (Injury, poisoning and procedural complications) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1
Impulse-control disorder (Psychiatric disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Amenorrhoea (Reproductive system and breast disorders) | 1/4 — The N for this adverse event has been adjusted to the number of females in the study as it is a sex-specific event.
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
The study was terminated by Alexion, as only 5 of the planned 12 participants were enrolled due to difficulty in recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-05-03): https://cdn.clinicaltrials.gov/large-docs/24/NCT04155424/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-15): https://cdn.clinicaltrials.gov/large-docs/24/NCT04155424/SAP_001.pdf